CLINICAL TRIAL: NCT02564198
Title: A Phase 1 Study Of Ramucirumab, a Human Monoclonal Antibody Against the Vascular Endothelial Growth Factor-2 (VEGFR-2) Receptor in Children With Refractory Solid Tumors, Including CNS Tumors
Brief Title: A Study of Ramucirumab (LY3009806) in Children With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15542; I4T-MC-JVDA (Other: Eli Lilly and Company); ADVL1416 (Other: Children's Oncology Group)
Record Dates: First submitted 2015-09-25; First posted 2015-09-30 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Pediatric Solid Tumor; Refractory Tumor; Recurrent Tumor; CNS Malignancies
Keywords: relapsed pediatric solid tumors; unspecified childhood solid tumor; brain and central nervous system tumors
MeSH Terms: conditions — Neoplasms; Recurrence; Central Nervous System Neoplasms | interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramucirumab (Experimental): (Part A-Non-CNS Solid Tumors) Escalating doses of 8 milligrams per kilogram (mg/kg) or 12 mg/kg Ramucirumab administered as an intravenous infusion every 2 weeks (Q2W) with 3 doses per 42 day cycle.
  (Part B-CNS Tumors) Participants received 12 mg/kg Ramucirumab as an intravenous injection Q2W with 3 doses per cycle.
  Interventions: Drug: Ramucirumab

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806; IMC-1121B; Cyramza

SUMMARY:
The main purpose of this study is to evaluate the safety of the study drug known as ramucirumab in children with recurrent or refractory solid tumors including central nervous system (CNS) tumors.

ELIGIBILITY:
Inclusion Criteria:

* Part A: participants with recurrent or refractory non-CNS solid tumors
* Part B: participants with recurrent or refractory CNS tumors
* Measurable or evaluable disease
* No other therapeutic options
* Performance Status: Karnofsky ≥50% for participants >16 years and Lansky ≥50 for participants ≤16 years

Exclusion Criteria:

* Active or recent history of serious bleeding events
* Active or recent history of gastrointestinal perforations, ulcers, fistulas or abscesses
* Active or recent history of hypertensive crisis or hypertensive encephalopathy
* Active non-healing wound or bone fracture
* History of solid organ transplant

Ages: 12 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2015-12-11 (Actual); Primary Completion 2019-07-16 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (21):
- United States (21):
  - Childrens Hospital of Alabama, Birmingham, Alabama
  - Children's Oncology Group, Monrovia, California
  - Childrens Hospital of Orange County, Orange, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Mark O Harfield-Warren Grant Magnuson Clinical Center, Bethesda, Maryland
  - University of Michigan Health Systems, Ann Arbor, Michigan
  - University of Minnesota Hospital, Minneapolis, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Childrens Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - St Jude Childrens Research Hospital, Memphis, Tennessee
  - Texas Childrens Hospital, Houston, Texas
  - Seattle Children's Hospital Research Foundation, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- See also: Click here for more information about this study: A Study of Ramucirumab (LY3009806) in Children With Refractory Solid Tumors — https://trials.lillytrialguide.com/en-US/trial/696R592JJCYO4i62eAqiSi

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers included participants who had progressive disease, death due to any cause or alive and on study at conclusion, but off treatment.
Groups:
- 8 mg/kg Ramucirumab (Part A): Participants received 8 milligram per kilogram [mg/kg] Ramucirumab administered as an intravenous infusion every 2 weeks (Q2W) with 3 doses per 42 day cycle.
- 12 mg/kg Ramucirumab (Part A); 12 mg/kg Ramucirumab (Part B): Participants received 12 mg/kg Ramucirumab as an intravenous injection Q2W with 3 doses per cycle.
Period: Overall Study
Arm/Group | 8 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part B)
Started | 8 | 15 | 6
Received at Least 1 Dose of Study Drug | 8 | 15 | 6
Completed | 6 | 10 | 6
Not Completed | 2 | 5 | 0
Not completed — Withdrawal by Subject | 2 | 4 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- 8 mg/kg Ramucirumab (Part A): Participants received 8 mg/kg Ramucirumab administered as an intravenous infusion Q2W with 3 doses per 42 day cycle.
- Total: Total of all reporting groups
Arm/Group | 8 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part B) | Total
Number analyzed (Participants) | 8 | 15 | 6 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.8 (3.33) | 11.9 (5.59) | 9.7 (5.9) | 12.5 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 2 | 12
  Male | 4 | 9 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 2 | 6
  Not Hispanic or Latino | 6 | 12 | 4 | 22
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 7 | 12 | 4 | 23
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 15 | 6 | 29

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Dose Limiting Toxicities (DLTs): Maximum Tolerated Dose of Ramucirumab
Description: A DLT is defined as an Adverse Event (AE) that is likely related to the study medication or combination, and fulfills any one of the following criteria, graded according to the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0:
  1. Any death not clearly due to the underlying disease or extraneous causes 2. Neutropenic fever 2. Any Grade ≥3 non-hematologic toxicity 3. Grade ≥4 neutropenia or thrombocytopenia >7 days 4. Grade ≥3 thrombocytopenia with bleeding 5. Grade ≥3 nausea/vomiting or diarrhea>72 hours with adequate antiemetic and other supportive care 6. Grade ≥3 fatigue ≥1 week 7. Grade ≥3 electrolyte abnormality that lasts>72 hours, unless the Participant has clinical symptoms, in which case all Grade 3+electrolyte abnormality regardless of duration should count as a DLT.
  8. Grade ≥3 prolongation of QT interval corrected using the Fridericia formula on 2 separate electrocardiogram readings approximately 5 min apart.
Time Frame: Baseline to Study Completion (Up to 42 Months)
Population: All randomized participants from Part A, who received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | 8 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part A)
Number analyzed (Participants) | 8 | 15
Participants | 1 | 1

2. Primary Outcome: Population Pharmacokinetics (PK): Minimum Concentration (Cmin) of Ramucirumab
Description: Population Pharmacokinetics (PK): Minimum observed plasma concentration of Ramucirumab.
Time Frame: Predose, Cycle 1 Day 1 (end of infusion (EOI), 1 hour after EOI) and Cycle 1 Day 43 (1 hour after EOI)
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data. Per protocol, 12 mg/kg Ramucirumab PK data were reported per dose level combining Part A and B participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Groups:
- 8 mg/kg Ramucirumab: Participants received 8 mg/kg Ramucirumab administered as an intravenous infusion every 2 weeks (Q2W) with 3 doses per 42 day cycle.
- 12 mg/kg Ramucirumab: Participants received 12 mg/kg Ramucirumab as an intravenous injection Q2W with 3 doses per cycle.
Arm/Group | 8 mg/kg Ramucirumab | 12 mg/kg Ramucirumab
Number analyzed (Participants) | 8 | 19
microgram per milliliter (µg/mL)
  Cycle 1 Day 1 | 30.0 (32) | 48.3 (41)
  Cycle 1 Day 43: number analyzed (Participants) | 4 | 16
  Cycle 1 Day 43 | 53.6 (31) | 80.2 (44)

3. Primary Outcome: Number of Participants With Anti-Ramucirumab Antibodies
Description: Number of participants with positive treatment emergent anti-ramucirumab antibodies was summarized by treatment group. A treatment-emergent anti-drug antibodies (TEADA) sample was defined as: a post treatment sample with at least a 4-fold increase in titer from pre treatment sample; or 1:20 post treatment titer for participants that had no detectable ADA titer at baseline.
Time Frame: Predose Cycle 1 Day 1 through Follow-Up (Up to 42 Months)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | 8 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part B)
Number analyzed (Participants) | 8 | 15 | 6
participants | 0 | 0 | 0

4. Secondary Outcome: Overall Response Rate (ORR): Percentage of Participants Who Achieve Complete Response (CR) or Partial Response (PR)
Description: Overall response rate is the best response of complete response (CR) or partial response (PR) as classified by the independent central review according to the Response Evaluation Criteria In Solid Tumors (RECIST v1.1). CR is a disappearance of all target and non-target lesions and normalization of tumor marker level. PR is an at least 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameter) without progression of non-target lesions or appearance of new lesions. Overall response rate is calculated as a total number of participants with CR or PR divided by the total number of participants per cohort with at least 1 measurable lesion, multiplied by 100. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline to Date of Objective Disease Progression (Up to 42 Months)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 8 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part B)
Number analyzed (Participants) | 8 | 15 | 6
Percentage of participants | 0 [0.0 to 41.0] | 0 [0.0 to 23.2] | 0 [0.0 to 45.9]

5. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR), Partial Response (PR) or Stable Disease (SD): Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) was the percentage of participants with a best overall response of CR, PR, or Stable Disease (SD) as per Response using RECIST v1.1 criteria. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. SD was neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD for target lesions, no progression of non-target lesions, and no appearance of new lesions. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Baseline to Date of Objective Disease Progression (Up to 42 Months)
Population: All randomized participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 8 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part B)
Number analyzed (Participants) | 8 | 15 | 6
Percentage of participants | 62.5 [29.0 to 96.3] | 40.0 [17.7 to 71.1] | 33.3 [4.3 to 77.7]

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR was the time from the date of first evidence of complete response or partial response to the date of objective progression or the date of death due to any cause, whichever is earlier. CR and PR were defined using the RECIST v1.1. CR defined as the disappearance of all target and non-target lesions and no appearance of new lesions. PR defined as at least a 30% decrease in the sum of the LD of target lesions (taking as reference the baseline sum LD), no progression of non-target lesions, and no appearance of new lesions. If a responder was not known to have died or have objective progression as of the data inclusion cutoff date, duration of response was censored at the last adequate tumor assessment date. PD was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions.
Time Frame: Date of Complete Response (CR) or Partial Response (PR) to Date of Objective Disease Progression or Death Due to Any Cause (Up to 42 Months)
Population: Zero participants analyzed. Duration of response was not evaluable, as there were no participants with CR or PR.
Arm/Group | 8 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part B)
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from date of randomization to the date of death (due to any cause). For participants whose last known status is alive at the data cutoff date for the analysis, time will be censored as the last contact date prior to the data cutoff date.
Time Frame: Baseline to Date of Death from Any Cause (Up to 42 Months)
Population: All randomized participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 8 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part B)
Number analyzed (Participants) | 8 | 15 | 6
Months | NA [NA to NA] — There were not enough events/deaths to compute a median or 95% confidence interval. | NA [NA to NA] — There were not enough events/deaths to compute a median or 95% confidence interval. | NA [NA to NA] — There were not enough events/deaths to compute a median or 95% confidence interval.

ADVERSE EVENTS:
Time Frame: Baseline, up to 4 years 8 months
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | 8 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part A) | 12 mg/kg Ramucirumab (Part B)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/15 | 0/6
Serious Adverse Events (participants affected / at risk) | 3/8 | 7/15 | 2/6
Other Adverse Events (participants affected / at risk) | 8/8 | 15/15 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 mg/kg Ramucirumab (Part A) (N=8) | 12 mg/kg Ramucirumab (Part A) (N=15) | 12 mg/kg Ramucirumab (Part B) (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 8 mg/kg Ramucirumab (Part A) (N=8) | 12 mg/kg Ramucirumab (Part A) (N=15) | 12 mg/kg Ramucirumab (Part B) (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 (4) | 9 (9) | 2 (3)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 5 (7) | 2 (3)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 5 (6) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (5) | 7 (7) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Tongue geographic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 7 (7) | 2 (3)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0)
Face oedema (General disorders) | 0 (0) | 2 (2) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 8 (9) | 1 (1)
Impaired healing (General disorders) | 1 (2) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 6 (6) | 1 (1)
Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 0 (0)
Coxsackie viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Post procedural discharge (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 6 (7) | 3 (3)
Anion gap increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 12 (14) | 2 (2)
Bacterial test positive (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 4 (5) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 2 (3) | 1 (2)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin increased (Investigations) | 1 (2) | 1 (6) | 3 (5)
International normalised ratio decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (7) | 2 (2) | 4 (5)
Neutrophil count decreased (Investigations) | 1 (2) | 5 (6) | 2 (2)
Platelet count decreased (Investigations) | 2 (3) | 3 (4) | 2 (3)
Prothrombin time shortened (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (5) | 1 (2)
White blood cell count decreased (Investigations) | 2 (2) | 6 (7) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 7 (9) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (8) | 1 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (4) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 3 (4)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (6) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 7 (7) | 2 (3)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 7 (12) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 2 (3)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (5) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 7 (8) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 2 (2) | 4 (4) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (4) | 6 (8) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (10) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 2 (2)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 6 (13) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 3 (8) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/98/NCT02564198/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT02564198/SAP_001.pdf